CLINICAL TRIAL: NCT06750237
Title: Effects of Balance Training Exercises Using Unstable and Stable Surfaces on Fall Risk Among Elderly Females
Brief Title: Effects of Balance Training Exercises Fall Risk Among Elderly Females
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0518
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Elderly Females
Keywords: Balance Training; stable; unstable; fall
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometrics (Experimental): will be an interventional group and will be treated by training the patients on unstable surfaces. The heating pad will be applied for 10 minutes as a warm-up. Then Isometric exercises of the lower limb and bridging for back extensors strengthening and improving patient confidence will be done. After that Single leg stance, Toe Raises, standing lower limb abduction and extension with proper support will be done and Mini Squats by stabilizing the patient against the wall or taking the help of an attendant or through a Stabilizing belt will be done. The session will last for 30 minutes. It will be conducted 2 months 3 times per week
  Interventions: Other: Unstable surface and isometrics
- Stable surface and isometrics (Active Comparator): will be an interventional group and will be treated by training the patients on stable surfaces. The heating pad will be applied for 10 minutes as a warm-up. Then Isometric exercises of the lower limb and bridging for back extensors strengthening and improving patient confidence will be done. After that Single leg stance, Toe Raises, standing lower limb abduction and extension with proper support will be done and Mini Squats by stabilizing the patient against the wall or taking the help of an attendant or through a Stabilizing belt will be done. The session will last for 30 minutes. It will be conducted 2 months 3 times per week.
  Interventions: Other: Stable surface and Isometrics

INTERVENTIONS:
Other: Stable surface and Isometrics — will be treated by training the patients on unstable surfaces. The heating pad will be applied for 10 minutes as a warm-up. Then Isometric exercises of the lower limb and bridging for back extensors strengthening and improving patient confidence will be done. After that Single leg stance, Toe Raises, standing lower limb abduction and extension with proper support will be done and Mini Squats by stabilizing the patient against the wall or taking the help of an attendant or through a Stabilizing belt will be done. The session will last for 30 minutes. It will be conducted 2 months 3 times per week
  Arms: Stable surface and isometrics
Other: Unstable surface and isometrics — and will be treated by training the patients on stable surfaces. The heating pad will be applied for 10 minutes as a warm-up. Then Isometric exercises of the lower limb and bridging for back extensors strengthening and improving patient confidence will be done. After that Single leg stance, Toe Raises, standing lower limb abduction and extension with proper support will be done and Mini Squats by stabilizing the patient against the wall or taking the help of an attendant or through a Stabilizing belt will be done. The session will last for 30 minutes. It will be conducted 2 months 3 times per week.
  Arms: Isometrics

SUMMARY:
Falls are the second leading cause of unintentional injury deaths globally, and the literature shows that 40% of community-dwelling older adults who are over 65 years old experience fall accidents annually. It also harms the well-being of the elderly, including the lack of access to daily services. Therefore, exercise interventions that target balance, gait, and muscle strength increase can effectively prevent falls in older adults.

A fall prevention program that includes strength and balance training and patient education can improve muscle balance and mental capacity in older women with a history of falls. dimensions of abilities of the elderly are improved by exercise, such as dynamic balance, static balance, participants fear of falling, balance confidence, quality of life, and physical performance. The study will be a randomized clinical trial and will be conducted in Fatima Memorial Hospital, and Atif Rehab Clinic. The sample size is calculated from the open epi tool. Considering the attrition rate (10%) the sample size is calculated to be 36 altogether. This study will be completed in a time duration of 10 months after the approval of the synopsis. Non-probability convenience sampling technique will be used and participants will be recruited in the study after randomization through the lottery method. The subjects will be divided into two groups. Baseline treatment is isometric of the lower limb and bridging. Group A will receive balance training exercises using unstable surfaces and Group B will receive balance training exercises using stable surfaces. The tools that will be used are the Fall Efficacy scale-international (FES-I), Berg Balance Scale ((BBS), and ABC (Activities-Specific Balance Coordination) Scale, and after data collection, data will be analyzed by using SPSS version 26.

ELIGIBILITY:
Inclusion Criteria

* Age between 60-75 years old (18)
* Sedentary lifestyle females
* No history of fracture and ligamentous injury in the last 6 months
* Muscular strength should be in at least Grade 3
* Berg Balance Scale score ≤ 49

Exclusion Criteria:

* Any chronic disease such as carcinoma
* Athletes
* Women underwent any surgery (hysterectomy) in the last 2 months

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-04-12 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Fall Efficacy Scale | baseline and fourth week
  Fall efficacy was measured by the Fall-Efficacy Scale-International (FES-I), a widely accepted tool for the evaluation of perceived confidence in performing a range of activities of daily living in the home and community environments, without falling (The FES-I contains 16 items, which are scored on a four-point scale. The scores range from 16 to 64 points, and higher scores indicate lower self-efficacy (20) The reliability of this tool is 0.94 and the validity is 0.84
Berg Balance Scale | baseline and fourth week
  The BBS is considered the "gold standard" for assessing balance, and it can evaluate dynamic and static balance functions simultaneously. It consists of 14 tasks of varying difficulty, and each item is scored on a scale of 0-4.31 The maximum score is 56, and higher scores indicate better performance. The reliability of this tool is 0.96
ABC (Activities-Specific Balance Coordination) Scale | baseline and fourthweek
  The scale includes 16 activities of daily living, such as walking around the house, sweeping the floor, and walking in a crowded mall, which needs complex posture control abilities (including posture stability and orientation) for adaptation to complex environments to maintain balance.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadaqa M, Nemeth Z, Makai A, Premusz V, Hock M. Effectiveness of exercise interventions on fall prevention in ambulatory community-dwelling older adults: a systematic review with narrative synthesis. Front Public Health. 2023 Aug 3;11:1209319. doi: 10.3389/fpubh.2023.1209319. eCollection 2023. PMID 37601180
- [Background] Sun M, Min L, Xu N, Huang L, Li X. The Effect of Exercise Intervention on Reducing the Fall Risk in Older Adults: A Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2021 Nov 29;18(23):12562. doi: 10.3390/ijerph182312562. PMID 34886293
- [Background] van Hoof J, Marston HR. Age-Friendly Cities and Communities: State of the Art and Future Perspectives. Int J Environ Res Public Health. 2021 Feb 9;18(4):1644. doi: 10.3390/ijerph18041644. PMID 33572181